CLINICAL TRIAL: NCT05191537
Title: Comparison of Spinal Mobilization With Arm Movement and Positional SNAGS on Pain and Disability in Cervical Radiculopathy Patients
Brief Title: Spinal Mobilization With Arm Movement and Positional SNAGS in Cervical Radiculopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0127 Maryam
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Radiculopathy, Cervical
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinal mobilization with arm movement (Experimental): conventional treatment and of spinal mobilization with arm movement
  Interventions: Other: shoulder Mobilization with arm movement
- positional SNAGs (Active Comparator): conventional treatment and positional SNAGs
  Interventions: Other: Sustained Natural Apophyseal Glides

INTERVENTIONS:
Other: Sustained Natural Apophyseal Glides — The patient sits well supported in a chair. The cervical spine and head are set in a neutral position. A painless passive posterior to anterior (PA) glide is applied in the plane of the facets on either the spinous process or the articular pillar/cervical lamina. While the glide is sustained the patient actively moves their neck in the direction that previously produced the symptoms. If symptom-free, the patient applies over-pressure further into the movement restriction. 3-6 repetitions are performed
  Arms: positional SNAGs
Other: shoulder Mobilization with arm movement — The patient is seated. The therapist contacts the length of the spinous process with the medial aspect of the thumb. A transverse glide is applied by the therapist's index finger against the thumb contacting the spinous process. The direction of the glide is to the contralateral side of the pain. While the mobilisation is sustained the patient moves their arm through a pain-free abduction range. 3-5 sets of 6-10 repetitions may be performed.
  Arms: spinal mobilization with arm movement

SUMMARY:
Data will be collected in Hussain Memorial Hospital by taking informed consent. Randomised clinical trial is conducted taking thirty patients of both genders with confirmed diagnoses of cervical radiculopathy, their ages ranged from 25 to 60. A cluster of winner to rule out patient with cervical radiculopathy. They will be randomly assigned into two groups by the lottery method. Group A will receive conventional treatment and of spinal mobilization with arm movement (intervention 1) Group B will receive conventional treatment and positional SNAGs (intervention 2). The treatment will be conducted at a frequency of three sessions per week for four weeks. Two values will be taken, one as baseline and the other at end of the session.

Then follow up the patient to rule out which intervention is more effective than the other. Neck Disability Index, Numeric Pain Rating Scale and ROM will be used to measure outcomes.

DETAILED DESCRIPTION:
the objective of the study is To compare the effect of spinal mobilization with arm movement and positional SNAGs on pain and disability in cervical radiculopathy patients.

The study design will be Randomized ClinicalTrial The sampling Technique will be Consecutive sampling technique

Tool:

The Neck Disability Index (NDI): used for measuring functional improvement in the neck.

Numeric Pain Rating Scale (NPRS): used for measuring pain.

Inclinometer: used for measuring Range of motion of cervical region.

Data will be collected in Hussain Memorial Hospital by taking informed consent. Randomised clinical trial is conducted taking thirty patients of both genders with confirmed diagnoses of cervical radiculopathy, their ages ranged from 25 to 60. A cluster of winner criteria will be used to rule out patient with cervical radiculopathy. They will be randomly assigned into two groups by the lottery method. Group A will receive conventional treatment and of spinal mobilization with arm movement (intervention 1) Group B will receive conventional treatment and positional SNAGs (intervention 2). The treatment will be conducted at a frequency of three sessions per week for four weeks. Two values will be taken, one as baseline and the other at end of the session.

Then follow up the patient to rule out which intervention is more effective than the other. Neck Disability Index, Numeric Pain Rating Scale and ROM will be used to measure outcomes.

ELIGIBILITY:
INCLUSION CRITERIA

* Symptoms duration more than 6 months.
* Age 25 -60
* The patient has confirm the diagnosis of Radiculopathy of cervical origin,
* VAS more than 5
* A cluster of Wainner 3 positive out of 4 EXCLUSION CRITERIA
* Malignancy
* Infection (such as osteomyelitis or diskettes)
* Osteoporosis
* Inflammatory arthritis
* Fracture
* Pregnancy
* Uncontrolled hypertension or cardiovascular disease
* Carotid or vertebral artery disease.
* Trauma cases

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 weeks.
  The numeric pain rating scale (NPRS) is a measurement scale that is used to measure a characteristic or attitude of pain. it is a 0-10 point scale. 0 mean no pain and 10 mean unbearable pain. Change from Baseline for pain Assessment at 4 weeks.
Neck Disability Index(NDI) | 4 weeks.
  NDI questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. It had 10 sections with total 50 scores. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage. 0 points or 0% means : no activity limitations , 50 points or 100% means complete activity limitation. Change from Baseline for disability Assessment at 4 weeks.
Inclinometer for range of motion | 4 weeks.
  It's a range measuring tool used for the Range of Motion of neck flexion, extension and rotation. If the angle increases its mean improving. Change from Baseline for Range of Motion Assessment at 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: muhammad sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- Hussain Memorial Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krivickas LS, Wilbourn AJ. Peripheral nerve injuries in athletes: a case series of over 200 injuries. Semin Neurol. 2000;20(2):225-32. doi: 10.1055/s-2000-9832. PMID 10946743
- [Background] Hee HT, Castro FP Jr, Majd ME, Holt RT, Myers L. Anterior/posterior lumbar fusion versus transforaminal lumbar interbody fusion: analysis of complications and predictive factors. J Spinal Disord. 2001 Dec;14(6):533-40. doi: 10.1097/00002517-200112000-00013. PMID 11723406
- [Background] Anandkumar S. The effect of sustained natural apophyseal glide (SNAG) combined with neurodynamics in the management of a patient with cervical radiculopathy: a case report. Physiother Theory Pract. 2015 Feb;31(2):140-5. doi: 10.3109/09593985.2014.971922. Epub 2014 Oct 20. PMID 25329587
- [Background] Shafique S, Ahmad S, Shakil-Ur-Rehman S. Effect of Mulligan spinal mobilization with arm movement along with neurodynamics and manual traction in cervical radiculopathy patients: A randomized controlled trial. J Pak Med Assoc. 2019 Nov;69(11):1601-1604. doi: 10.5455/JPMA.297956.. PMID 31740863